CLINICAL TRIAL: NCT00930631
Title: Pharmacokinetics, Metabolism and Elimination of Tritiated [3H] BMS747158 in Healthy Male Subjects
Brief Title: Study of [3H] BMS747158 in Healthy Male Subjects
Acronym: PPA103
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BMS747158-103
Record Dates: First submitted 2009-06-24; First posted 2009-06-30 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2011-10

CONDITIONS: Coronary Artery Disease
Keywords: CAD; Pharmacokinetics; BMS747158
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): Single arm PK study
  Interventions: Drug: [3H] BMS747158

INTERVENTIONS:
Drug: [3H] BMS747158 — Single bolus intravenous injection of [3H] BMS747158

SUMMARY:
The purpose of this clinical study is to assess the safety, extent and route of [3H] BMS747158 radioactivity eliminated (mass balance) in urine and feces of healthy male subjects. The safety of [3H] BMS747158 administration will also be assessed, as well as pharmacokinetics of [3H] BMS747158 and metabolite identification.

DETAILED DESCRIPTION:
This Phase I, nonrandomized, open-label study will enroll up to seven healthy male subjects who meet all of the inclusion and none of the exclusion criteria. Subjects will receive 100 (±20) μCi of [3H] BMS747158. Subjects will undergo blood, urine, and fecal collections to evaluate [3H] activity for a minimum of 7 days post-dose. Safety will be assessed by monitoring of adverse events (AEs), vital signs, physical examinations, clinical laboratory tests, and electrocardiograms (ECGs).This Phase I, nonrandomized, open-label study will enroll up to seven healthy male subjects who meet all of the inclusion and none of the exclusion criteria. Subjects will receive 100 (±20) μCi of [3H] BMS747158. Subjects will undergo blood, urine, and fecal collections to evaluate [3H] activity for a minimum of 7 days post-dose. Safety will be assessed by monitoring of adverse events (AEs), vital signs, physical examinations, clinical laboratory tests, and electrocardiograms (ECGs).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written signed informed consent prior to any study procedures
2. Be healthy as determined by no clinically significant deviation from normal in medical history, physical examination, vital signs, ECG, and clinical laboratory tests
3. Have a Body Mass Index (BMI) of 18 to 30 kg/m2
4. Be male, age 18 to 45 years
5. Be sterile or agree to use from admission until discharge one of the following approved methods of contraception:

   * a male condom with spermicide
   * a sterile sexual partner
   * use by female sexual partner of an intrauterine device (IUD) with spermicide *a female condom with spermicide contraceptive sponge with spermicide
   * an intravaginal system [e.g., NuvaRing®]
   * a diaphragm with spermicide
   * a cervical cap with spermicide, or
   * oral, implantable, transdermal, or injectable contraceptives
6. Must be able to communicate effectively with study personnel

Exclusion Criteria:

1. Any significant active or chronic medical illness or acute significant trauma
2. History of any condition that may disrupt and/or increase permeability of the blood-brain barrier or diabetes
3. History of any neurological disease.
4. History of concussion or meningitis within the past 6 months
5. History of sleep disorders, including snoring with sleep apnea and narcolepsy
6. History of anxiety disorder
7. Current or recent GI disease
8. Major surgery within 4 weeks
9. GI surgery that could impact upon the re-absorption of study drug
10. History of chronic constipation
11. History of asthma as deemed clinically significant by the Investigator or designee
12. History of recent (within 2 weeks of enrollment) infection (e.g., upper respiratory tract infection, urinary tract infection)
13. Known and confirmed drug allergies or hypersensitivities
14. Donation of blood and/or plasma to a blood bank or in a clinical study (except as required for screening) within four weeks of enrollment
15. Blood transfusion within four weeks of enrollment
16. Inability to tolerate intravenous medication or unlikely to obtain and/or tolerate venous access
17. Past (6 months) or present history of drug or alcohol abuse
18. Screening or pre-dose ECG interval abnormalities or organ dysfunction.
19. Positive urine screen for drugs of abuse either at screening or before dosing
20. Positive blood screen for hepatitis B surface antigen, hepatitis C antibody, or HIV
21. Exposure to any investigational drug, device, or placebo within four weeks of enrollment
22. Use of any prescription drugs within 4 weeks of enrollment
23. Use of any other drugs, including over-the-counter medications (e.g., acid-controllers) and herbal preparations within two weeks of enrollment
24. Smoking within 1 month of enrollment
25. Alcohol or caffeine consumption within 72 hours of study drug administration
26. Participation in a radio-labeled study within 12 months of enrollment
27. Intake of radio-labeled drug substance or exposure to significant radiation
28. Participation in any prior study with BMS747158

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To assess safety and the extent and route of [3H] radioactivity eliminated (mass balance) in urine and feces following a single intravenous (IV) dose of approximately 100 (±20) µCi of [3H] BMS747158 in healthy male subjects. | August 2009

SECONDARY OUTCOMES:
To assess the pharmacokinetics (PK) of [3H] radioactivity and of [3H] BMS747158 in blood. To identify the major metabolites of [3H] BMS747158 present in blood, urine, and feces | August 2009

CONTACTS AND LOCATIONS:
Overall Officials: Debra A Mandarino, MD, Principal Investigator — Covance Clinical Laboratory Unit
Locations (1):
- Covance Clinical Laboratory Unit, Madison, Wisconsin, United States